CLINICAL TRIAL: NCT06415682
Title: The Efficacy and Mechanism of SMA+M1 Repetitive Transcranial Magnetic Stimulation on Freezing of Gait in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-SR-290
Record Dates: First submitted 2024-05-05; First posted 2024-05-16 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; gait symptoms; freezing of gait; TMS; neural mechanism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- double-site high frequency rTMS over the bilateral M1 of the lower leg and SMA (Experimental): Patients in the Experimental group underwent ten sessions of double-site high frequency rTMS over the bilateral M1 of the lower leg and SMA.
  Interventions: Device: SMA+M1 Transcranial Magnetic Stimulation
- single-site high frequency rTMS over the bilateral M1 of the lower leg (Active Comparator): Patients in the Active Comparator group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral M1 of the lower leg.
  Interventions: Device: M1 Transcranial Magnetic Stimulation
- sham magnetic stimulation on the bilateral M1 of the lower leg (Sham Comparator): Patients in the Sham Comparator group underwent ten sessions of double sham rTMS on the bilateral M1 of the lower leg.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: SMA+M1 Transcranial Magnetic Stimulation — The M1 stimulation session consisted 40 trains of 10-Hz rTMS with the protocol of 5s train session and 25s intertrain intervals. There were 4000 pulses per day for M1-LL (unilateral stimulation 2000 pulses). For SMA stimulation, a 5s burst of 10Hz rTMS was repeated 20 times (1000 pulse, 20 minutes' duration).
  Patients in the Experimental group underwent ten sessions of double-site high frequency rTMS over the bilateral primary motor cortex (M1) of the lower leg and supplementary motor area (SMA).
  Arms: double-site high frequency rTMS over the bilateral M1 of the lower leg and SMA
Device: M1 Transcranial Magnetic Stimulation — The M1 stimulation session consisted 40 trains of 10-Hz rTMS with the protocol of 5s train session and 25s intertrain intervals. There were 4000 pulses per day for M1-LL (unilateral stimulation 2000 pulses). Patients in the Active Comparator group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral M1 of the lower leg.
  Arms: single-site high frequency rTMS over the bilateral M1 of the lower leg
Device: Sham Transcranial Magnetic Stimulation — Patients in the Sham Comparator group underwent 10 sessions of double sham rTMS on M1 of the lower leg.
  Arms: sham magnetic stimulation on the bilateral M1 of the lower leg

SUMMARY:
This study is a double-blinded randomized study examining the efficacy of the double-site (M1+SMA) repetitive transcranial magnetic stimulation on Freezing of Gait (FOG) in patients with Parkinson's disease. The investigators hypothesize that treatment using magnetic stimulation on double site (including M1-LL and SMA) will improve FOG and gait symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Patients in the double-site group underwent ten sessions of double-site high frequency rTMS over the bilateral primary motor cortex of the lower leg and supplementary motor area, whereas patients in the single-site group underwent ten sessions of single-site active magnetic stimulation with high frequency rTMS over the bilateral primary motor cortex of the lower leg. In addition, patients in the sham group underwent 10 sessions of sham rTMS on bilateral primary motor cortex of the lower leg. Assessments of FOG severity, gait, motor symptoms, excitability of cortex motor (using transcranial magnetic stimulation), plasma indicators and multimodal magnetic resonance were performed three times: at baseline, one day post intervention, one month post intervention.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 40-80 years;
2. diagnosis of idiopathic Parkinson's disease (PD) according to the Movement Disorder Society clinical diagnostic criteria;
3. patients were stable on dopaminergic treatment for at least 3 months;
4. Item 3 of the Freezing of Gait Questionnaire(FOG-Q) scored ≥1;
5. Patients experienced FOG during an interview.

Exclusion Criteria:

1. comorbidities of major neurologic diseases other than PD;
2. suffer from musculoskeletal disorders that could have interfered with their ability to walk;
3. presence of contraindications for transcranial magnetic stimulation (TMS) and magnetic resonance imaging (MRI);
4. marked tremor interfered with TMS detection;
5. previously receiving any kinds of TMS interventions;
6. severe cognitive impairment making cooperation impossible [Mini Mental State Examination (MMSE) < 24];
7. were unable to walk independently during the OFF state.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Changes of Freezing of Gait severity | Assessed at baseline, one day post intervention, one month post intervention
  The Freezing of Gait questionnaire will be used to quantify the frequency and severity of FOG. The score will be compared to the baseline. The minimum and maximum values of the FOGQ are 0 and 24. A higher score means a worse outcome. The differences in FOGQ scores before and after treatment can be used to evaluate the effect of TMS treatment.

SECONDARY OUTCOMES:
Freezing of Gait severity assessment | Assessed at baseline, one day post intervention, one month post intervention
  The New Freezing of Gait questionnaire will be used to quantify the frequency and severity of FOG. The score will be compared to the baseline. The minimum and maximum values of the NFOGQ are 0 and 28. A higher score means a worse outcome. The differences in NFOGQ scores before and after treatment can be used to evaluate the effect of TMS treatment.
Changes of Movement Disorder Society Unified Parkinson's disease rating scale part III (MDS-UPDRS-III) | Assessed at baseline, one day post intervention, one month post intervention
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms and non-motor symptoms. The minimum value is 0 and the maximum value is 132. A higher score means a worse outcome. The score will be compared to the baseline. The differences in MDS-UPDRS III part scores before and after treatment can be used to evaluate the effect of TMS treatment.
Changes of Gait speed | Assessed at baseline, one day post intervention, one month post intervention
  Gait speed (m/s) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in gait speed before and after treatment can be used to evaluate the effect of TMS treatment.
Changes of Stride length | Assessed at baseline, one day post intervention, one month post intervention
  Stride length (cm) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test. The differences in stride length before and after treatment can be used to evaluate the effect of TMS treatment.
Changes in Short-interval intracortical inhibition (SICI), intracortical facilitation (ICF) and short-interval intracortical facilitation (SICF) | Assessed at baseline, one day post intervention
  Short-interval intracortical inhibition (SICI), intracortical facilitation (ICF) and short-interval intracortical facilitation (SICF) are conducted by TMS devices to assess the cortical excitation and inhibition. SICI was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with 2ms, 3ms, 4ms interstimulus interval between conditioning and test stimuli. ICF was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with 10, 12, 15 ms interstimulus interval between conditioning and test stimuli. For SICF, a subthreshold first stimulus (S1) intensity was set at 1 mV and a subsequent suprathreshold second stimulus (S2) intensity was set at RMT. Interstimulus intervals were 1.0 to 5.0 milliseconds with increments of 0.5 millisecond.The differences in SICI, ICF and SICF before and after treatment can be used to evaluate the effect of TMS treatment.
Changes in functional connectivity in the brain cortex | Assessed at baseline, one day post intervention
  The functional connectivity in the brain cortex will be recorded by functional MRI. The differences in brain regions' functional connectivity before and after treatment can be used to evaluate the effect of TMS treatment.
Changes in brain structure | Assessed at baseline, one day post intervention
  Studying the brain structure among groups. The differences in brain microstructure before and after treatment can be used to evaluate the effect of TMS treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No